CLINICAL TRIAL: NCT05938205
Title: Multicomponent Analysis of phYsical Frailty BiomarkErs: Focus on Mitochondrial Health - MAYBE
Acronym: MAYBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: Università degli Studi di Brescia (Other); Azienda Ospedaliera di Padova (Other); University of Milan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1956CESC
Record Dates: First submitted 2020-02-21; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Sarcopenic Obesity; Frailty; Malnutrition; Protein
MeSH Terms: conditions — Frailty; Kwashiorkor

STUDY DESIGN:
Intervention Model Description: Single-center open-label randomized experimental study with 3 parallel arms with an allocation ratio of 1:1:1. Participants will be all involved in high intensity exercise (Exe-H). Participants will be further randomized into 3 groups to receive (double-blind) dietary supplementation with either placebo, low dose amino acid blend (AA-1) or full dose amino acid blend (AA-2).
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exe-H + placebo (Experimental): high intensity physical exercise combined with placebo
  Interventions: Behavioral: Placebo; Behavioral: Exe-H
- Exe-H + AA-1 (Experimental): high intensity physical exercise combined with low dose of aminoacids
  Interventions: Dietary Supplement: AA-1; Behavioral: Exe-H
- Exe-H + AA-2 (Experimental): high intensity physical exercise combined with high dose of aminoacids
  Interventions: Dietary Supplement: AA-2; Behavioral: Exe-H

INTERVENTIONS:
Dietary Supplement: AA-1 — low dose aminoacids
  Arms: Exe-H + AA-1
Dietary Supplement: AA-2 — high dose aminoacids
  Arms: Exe-H + AA-2
Behavioral: Placebo — Nutritional Placebo
  Arms: Exe-H + placebo
Behavioral: Exe-H — high intensity physical exercise

SUMMARY:
The study will be conducted in a group of obese sarcopenic patients (Sarco-Ob) aged > 60 years on moderately hypocaloric diet therapy aimed at comparing the effect of a strength exercise protocol, combined or not with dietary supplementation with amino acids, on physical performance, muscle strength, body composition, muscle oxidative metabolism, and biomarkers of sarcopenia. The supplementation study will be conducted in a double-blind manner.

DETAILED DESCRIPTION:
In this double-blind randomised control trial, older men, and women resident in Verona (Italy) will be selected from the Geriatrics Nutritional Clinic of the Borgo Trento Hospital or were contacted by telephone. A specific medical screening was initially programmed to verify the criteria of recruitment.

Anthropometric and body composition In the morning, in a fasted state, body mass will be taken with an electronic scale (Tanita electronic scale BWB-800 MA) and stature will be measured with a Harpenden stadiometer (Holtain Ltd., Crymych, Pembs. UK); BMI will be calculated as weight (kg)/height (m)2. Thereafter, total and regional body composition will be evaluated by means of dual-energy X-ray absorptiometry (DXA) using a total body scanner (QDR Horizon W, Hologic, MA, USA; fan-bean technology, software for Windows XP version 12.4.2) according to the manufacturer's procedures. Furthermore, the ALMI will be calculated as the sum of lean mass of arms and legs divided by height squared.

Physical performance On the same day, the SPPB test will be used to assess functional performance of the lower extremities. Each participant will performed: 4 m at usual customary gait speed, a five repeated chair-stands test and three standing balance tests (side by side, semi-tandem and tandem).

A digital dynamometer (CAMRY, Digital Hand Dynamometer model: EH101) will be used to assess HGS and all measurements were conducted by the same operator. Before starting, participants will observe a demonstration of the test procedure and engage in two practice attempts.

Knee muscle strength measurements and analysis An isokinetic dynamometer (CMSi Cybex Humac Norm Dynamometer, Lumex, Ronkokoma, NY, USA) will be used to assess the isokinetic strength of knee flexors and extensors muscles.

Maximal isokinetic knee extension-flexion tests will be performed in a randomised sequence at 60, 90, 150, 180 and 210°ˑs-1. Trials will consist in three knee extension-flexion movements with 60 s-recovery. The maximal strength of knee extensors muscle will be calculated with the Hill's hyperbolic function. The isokinetic knee extension-flexion power will be calculated as the product between strength and velocity. Finally, for knee extensors, maximal muscle power expressed in Watt, will be calculated from the power-velocity curve.

1-RM assessment Before starting training intervention, participants will perform three sessions of familiarization with the resistance isotonic machines. High intensity strength exercise (Exe-H) protocol: All the participants will performed a supervised progressive resistance training protocol, three times per week, 1 hour per session. Each participant will performed the same strength training protocol, starting with 3 sets of 8-10 repetitions at 70% of 1-RM (month 1), with a progressive increase of intensity at 75% of 1-RM (month 2 and month 3), and 80% 1-RM that will be maintained for the rest period of intervention. The compliance will be define as the number of exercise sessions expressed in % of the target value. Each participant will must reach a compliance above the 70% to be included in the final analysis.

ELIGIBILITY:
Inclusion Criteria:

Participants will be included in the study based on the following inclusion criteria:

* Older men and women between 60-80 years
* The presence of sarcopenic obesity was considered when the following two conditions were satisfied: Fat mass > 34.8% and FFM <90% of subject's ideal FFM.
* Resident in Verona (Italy)
* Stable weight in the previous 2 months
* Previously sedentary (less than one hour of exercise per week in the last 6 months)
* Signing of the informed consent for participation in the study

Exclusion criteria:

* Unstable angina or recent myocardial infarction
* Malignant or unstable arrhythmias
* Heart failure NYHA class > II
* Severe respiratory failure
* Severe heart valve disease (i.e severe aortic stenosis or insufficiency)
* Abdominal and/or thoracic aneurysm
* Recent intracerebral or subdural haemorrhage
* Poorly controlled arterial hypertension
* Presence of pacemakers or metal prostheses
* Severe chronic renal failure
* Symptomatic musculoskeletal pathology
* Symptomatic disc herniation, arthrosis, acute joint, tendon and ligamentous injuries, hip and/or knee prostheses recently placed (<6 months) or with joint instability, symptomatic or large inguinal or abdominal hernia
* Acute retinal detachment or bleeding
* Recent eye surgery (laser, cataract, retinal surgery, glaucoma surgery)
* History of malignant cancer within the previous 5 years
* Diagnosis of dementia
* Eating disorders

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline 1-repetition maximum with isokinetic dynamometer at 5-months | Month0, Month5
  Change in 1-repetition maximum test performed with isokinetic dynamometer in Kilograms

SECONDARY OUTCOMES:
Change from baseline Short Physical Performance Battery at 5-months | Month0, Month 5
  Change in Short Physical Performance Battery Score
Change from baseline in handgrip at 5-months | Month0, Month5
  Change in upper limb muscle strength measured with handgrip in kilograms
Changesfrom baseline skeletal muscle mass at 5-months | Month0, Month5
  Change skeletal muscle mass measured with DXA in kilograms
Change from baseline fat mass at 5-months | Month0, Month5
  Change fat mass measured with DXA in kilograms
Change from baseline in mRNA at 5-months | Month0, Month5
  Change mRNA dosage
Change from baseline in muscle power at 5-months | Month0, Month5
  Change in isokinetic muscle power of the lower limbs in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Elena Zoico, PhD, Study Director — Universita di Verona
Locations (1):
- AOUI Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Healthy Aging Center Verona web site — https://www.aovr.veneto.it/web/healthyaging/chi-siamo